CLINICAL TRIAL: NCT05330143
Title: A Phase II Multi-center, Randomized, Blind, Placebo-controlled Study to Evaluate Safety, Tolerance and Efficacy of ASC22 Combined With ART in Subjects With Human Immunodeficiency Virus
Brief Title: Study to Evaluate Safety, Tolerance and Efficacy of ASC22 Combined With ART in Subjects With HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASC22-204
Record Dates: First submitted 2022-03-17; First posted 2022-04-15 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: HIV-1-infection; HIV Infections; PD-L1 Gene Mutation
Keywords: ASC22; HIV; PD-L1
MeSH Terms: conditions — HIV Infections | interventions — envafolimab; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASC22 1mg/kg (Experimental): ASC22 Injection of 1mg/kg and anti-retroviral therapy for 12 weeks
  Interventions: Drug: ASC22 1mg/kg; Drug: Antiretroviral Therapy
- ASC22 2.5mg/kg (Experimental): ASC22 Injection of 2.5mg/kg and anti-retroviral therapy for 12 weeks
  Interventions: Drug: ASC22 2.5mg/kg; Drug: Antiretroviral Therapy
- Placebo (Placebo Comparator): 0.9% Saline and anti-retroviral therapy for 12 weeks
  Interventions: Drug: Antiretroviral Therapy; Drug: Placebo

INTERVENTIONS:
Drug: ASC22 1mg/kg — ASC22 single-dose of 1mg/kg vials administered subcutaneously once 4 week.
  Other Names: KN035
  Arms: ASC22 1mg/kg
Drug: ASC22 2.5mg/kg — ASC22 single-dose of 2.5mg/kg vials administered subcutaneously once 4 week.
  Other Names: KN035
  Arms: ASC22 2.5mg/kg
Drug: Antiretroviral Therapy — standard antiretroviral therapy including Integrase inhibitors (INSTIs)
Drug: Placebo — 0.9% saline vials administered subcutaneously once 4 week.
  Arms: Placebo

SUMMARY:
This study is a phase II, multicenter, randomized, blind, placebo-controlled to evaluate the safety, tolerance, efficacy of ASC22 injection in combination with anti-retroviral therapy to treat subjects living with human immunodeficiency virus type 1.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤ 60 years old at screening.
* Treated with anti-retroviral medicine continuously for at least 12 months within 6 months of diagnosis of HIV-1 infection.
* Treated with anti-retroviral medicine continuously, contain integrase inhibitor, for at least months before screening.
* CD4+ Cell count ≥300 cells/μL and CD4+/ CD8+ratio ≤ 0.9 at screening.
* Weight ≥ 50 kg at screening.

Exclusion Criteria:

* Known allergy to the drug or excipients used in this trial.
* HIV-associated opportunistic infections in the past 5 years.
* Co-sensors of HBV, HCV, syphilis, etc.
* With bleeding disorders or on anticoagulant therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
CD4/CD8 ratio changes compared with baseline | Week 4\Week 8\Week 12

SECONDARY OUTCOMES:
HIV-DNA copy changes compared with baselnie | Week 12
CD4+ count changes compared with baseline | Week 12
CD8+ count changes compared with baseline | Week 12
HLA-DR number changes compared with baseline | Week 12
CD38 count changes compared with baseline | Week 12
IL-2 concentration changes compared with baseline | Week 4\Week 8\Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Medical Center of the General Hospital of the Peoples Liberation Army, Beijing, Beijing Municipality, China